CLINICAL TRIAL: NCT05140031
Title: Keeping It Simple - Implementing Pain Education for All: a Clinical Cross-over Feasibility Study Among Chronic Pain Patients Referred to Community-based Rehabilitation
Brief Title: Keeping It Simple - Implementing Pain Education for All
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Municipality of Koege, Denmark (Unknown); Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Christian Lund Straszek, Ms.c, Ph.d. student, Aalborg University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Keeping it simple
Record Dates: First submitted 2021-11-06; First posted 2021-12-01 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: After a period of "usual care" for 2-4 weeks, we want to cross-over and add the pain education intervention.
  The pain education intervention is an add-on to "usual care" and consists of an individualized pain education program in the form of Danish PNE4Adults. The education program consists of two session of +/- 1 hour each tailored individually to the needs of the patient. After the pain education, the patient will continue the planned rehabilitation program, but will integrate the knowledge obtained through the pain education, as an integrated part of the PNE4Adults program.
Masking Description: This study is designed as a cross-over study. As such, all participants will receive usual care before being introduced to the PNE4Adults board.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Participants will initially undergo 2 weeks of usual care.
  Interventions: Other: PNE4Adults
- PNE4Adults (Experimental): Participants will undergo 2 sessions (1-2 weeks) where they will be introduced to the PNE4Adult board.
  Interventions: Other: PNE4Adults

INTERVENTIONS:
Other: PNE4Adults — It is a clear and concise program, that consists of a manual for the physiotherapist delivering the education and a board game to enhance engagement and participant involvement. It not only provides the physiotherapist with a clear "how-to" manual but also provides an easy and accessible way for the patient to grasp the difficult and complex concept of pain.

SUMMARY:
Pain education has proven difficult to implement into clinical practice. In Denmark 4 out of 10 adults has inadequate health literacy levels. To avoid inequality in health care we need a new and accurate method to provide pain education to all who need it.

In this study, existing concept of pain education is implemented into clinical practice for a group of chronic pain patients including those with low degrees of health literacy, and then evaluate its use from both patient and physiotherapist perspective.

DETAILED DESCRIPTION:
The focus of this is project is to implement existing knowledge into clinical practice and to adapt and test a tool (i.e., PNE4Kids) that was initially developed to explain pain to children and their parents, for its potential to teach adults in pain about contemporary pain science in a way that takes into consideration those with low degrees of health literacy. Further, we want to test its feasibility in adult pain patients at a community-based rehabilitation center. It is expected that adult patients suffering from chronic pain will find the adapted PNE4Kids, named PNE4Adults, comprehendible, will benefit from this type of pain education in terms of increased pain knowledge and self-efficacy, and decreased pain-intensity and pain catastrophizing thoughts. It is also expected that physiotherapists will find the pain education program easy to engage with and to transfer into a clinical setting.

ELIGIBILITY:
Eligible patients are; Danish speaking adult patients (≥18 years) Patients with chronic musculoskeletal pain (pain ≥ 3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of the PNE4Adults | During the final consultation, after approximeatly 6 weeks
  Acceptability of the combined intervention of PNE4Adults and usual care will be measured by a participant acceptability questionnaire on a 7-point Likert scale ranging from "very unacceptable", "unacceptable", "slightly unacceptable", "neither unacceptable nor acceptable", "slightly acceptable", "acceptable", and "very acceptable".
Comprehensibility of the PNE4Adults | During the final consultation, after approximeatly 6 weeks
  How comprehensible the PNE4Adults is, will be measured by a participant questionnaire on a 7-point Likert scale ranging from "very incomprehensible", "comprehensible", "slightly incomprehensible", "neither incomprehensible nor comprehensible", "slightly comprehensible", "comprehensible", and "very comprehensible".

SECONDARY OUTCOMES:
Concept of Pain Inventory (COPI-adult) | T0: Baseline, T1: at 2-3 weeks of usual care, T2: at one week after two sessions of PNE4Adults, T3: at additional 2-3 weeks of usual care
  To assess adults' beliefs and knowledge of pain science, a Danish version of the Concept of Pain Inventory (COPI-adult) is used. It is a 13-item self-reported questionnaire with the following response options; "strongly disagree", "disagree", "unsure", "agree", "strongly agree".
Pain Self-Efficacy scale, | T0: Baseline, T1: at 2-3 weeks of usual care, T2: at one week after two sessions of PNE4Adults, T3: at additional 2-3 weeks of usual care
  A questionnaire which measures how confident a person feels in dealing with everyday life despite having chronic pain. The PSEQ consists of 10 items, rated on a 7-point Likert scale ranging from 0 ("not confident at all") to 6 ("very confident").
Pain intensity | T0: Baseline, T1: at 2-3 weeks of usual care, T2: at one week after two sessions of PNE4Adults, T3: at additional 2-3 weeks of usual care
  Pain intensity is assessed on Numeric Rating Scale (NRS) with answer options ranging from 0 = ("no pain") to 10 = ("worst imaginable pain"). We will collect average pain intensity last 24 hours (NRSavg), worst pain intensity last 24 hours (NRSmax) and current pain intensity (NRScur) as they all seem to convey different aspects of pain and together provide a more accurate measure of pain.
Pain Catastrophizing Scale | T0: Baseline, T1: at 2-3 weeks of usual care, T2: at one week after two sessions of PNE4Adults, T3: at additional 2-3 weeks of usual care
  A questionnaire to assess catastrophizing in relation to actual or anticipated pain. The questionnaire has 3 sub-scales (i.e., rumination, magnification, and helplessness) and contains a total of 13-items. Patients use the same 5-point Likert-scale to respond to all 13 items ranging from "not at all" to "very much so"

CONTACTS AND LOCATIONS:
Locations (1):
- Køge Kommune, Køge, Region Zeland, Denmark

IPD SHARING:
Plan to Share IPD: No